CLINICAL TRIAL: NCT06581367
Title: Tailoring Antibiotic Duration for Respiratory Tract Infections in Primary Care: a Pragmatic Randomized Controlled Trial
Brief Title: Tailoring Antibiotic Duration for Respiratory Tract Infections in Primary Care
Acronym: STORM
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IJG-STORM-2024
Record Dates: First submitted 2024-08-28; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Acute Respiratory Tract Infection
Keywords: Antibacterial Agents Antimicrobial Resistance; Duration; Primary Health Care; Personalized Medicine; Drugs, Customized; Drug Resistance, Microbial; Patient-Centered Care

STUDY DESIGN:
Intervention Model Description: Patients with acute RTIs will be randomized to either usual care (full-course antibiotic therapy based on current guidelines), or a tailored approach (patients will be advised to visit the center as soon as they feel better and are afebrile for a clinical assessment and C-reactive protein rapid testing after completing two full days of antibiotic).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): Full-course antibiotic therapy based on current guidelines (7 days).
  Interventions: Drug: Complete a 7-day course
- Intervention group (Active Comparator): In the intervention group, patients will be advised to visit the center as soon as they feel better and are afebrile for a clinical assessment and C-reactive protein rapid testing after completing two full days of antibiotic.
  Interventions: Drug: Tailoring the course duration to the patient's needs.

INTERVENTIONS:
Drug: Tailoring the course duration to the patient's needs. — Patients will be advised to visit the center as soon as they feel better and are afebrile for a clinical assessment including vital signs (temperature, blood pressure, respiratory rate, pulse, and oxygen saturation) and C-reactive protein rapid testing after completing two full days of antibiotic.
  Other Names: Patient-centered approach
  Arms: Intervention group
Drug: Complete a 7-day course — The antibiotic course must be completed (7 days at least).
  Other Names: Completion of the antibiotic course
  Arms: Control group

SUMMARY:
The rise of drug-resistant organisms and the need to minimize side effects calls for a new approach to antibiotic therapy duration. This study explores tailoring the length of antibiotic treatment to patient recovery, focusing on whether adjusting therapy based on when the patient feels better is as effective as completing the prescribed course for acute respiratory tract infections (RTIs). The investigators will enroll 474 outpatients aged 18-75 with acute RTIs across 25 Spanish healthcare centers. Patients will be randomized into two groups: one following standard full-course antibiotic therapy, and another receiving a tailored approach, where treatment may be shortened based on clinical assessments. The primary outcome is clinical efficacy at day 14. Secondary outcomes include antibiotic duration, complications, and quality of life.

DETAILED DESCRIPTION:
Background. Combating the rise of drug-resistant organisms and minimizing the side effects demand a shift in how we approach antibiotic therapy duration. A study focused on tailoring antibiotic length of therapy to patients' needs as soon as they feel better, is a promising strategy. The investigators aim to assess whether adjusting the duration of antibiotic therapy according to individual patient needs, shortening it to the time when the patient feels better, proves as effective as completing the antibiotic course in acute respiratory tract infections (RTIs).

Methods. The investigators plan to enroll a minimum of 474 outpatients ranging from 18 to 75 years of age with clinical features of acute RTIs across 25 Spanish primary healthcare centers. Patients diagnosed with acute lower RTIs or acute rhinosinusitis, deemed by clinicians to require a beta-lactam course, will be randomized to either usual care, involving a full-course antibiotic therapy based on current guidelines, or a tailored approach. In the intervention group, patients will be advised to visit the center as soon as they feel better and are afebrile for a clinical assessment and C-reactive protein rapid testing after completing two full days of antibiotic. Treatment will be discontinued if these clinical results are normal. The primary outcome will be overall clinical efficacy at day 14, while secondary outcomes include duration, doses of antibiotic taken, complications and reattendance within the first month, drug-related adverse events, antibiotic given, other therapies, days of severe and moderate symptoms, days of symptoms, absenteeism and health-related quality of life. All participants will be given a symptom diary, recording their symptoms each evening. Additionally, a cost-effectiveness study and qualitative studies involving clinicians and patients aimed at exploring the strategy's pros, cons, uptake, and satisfaction levels will be carried out.

Discussion. The investigators will examine whether adults who present with symptoms of acute lower RTI or rhinosinusitis in general practice, who are treated with antibiotic courses until they feel better are as effective as longer standard courses. It is highly important that a possible reduction in the antibiotic course as soon as the patient feels better does not compromise patients' recovery or clinical course, which we will assess closely. This comprehensive approach aims to shed light on the practicality and impact of tailoring antibiotic duration in RTIs.

ELIGIBILITY:
Inclusion Criteria:

* Either adults with a) acute cough (new cough or worsening of a previous cough) as the predominant symptom which the clinician believes to be a bacterial acute lower RTI, such as community-acquired pneumonia, acute bronchitis or acute chronic obstructive pulmonary disease (COPD) exacerbations, or b) an acute bacterial rhinosinusitis
* Doctors deem beta-lactam therapy (given every eight hours for a minimum of seven days) is necessary

Exclusion Criteria:

* RTIs different from a lower RTI or acute rhinosinusitis
* Patients with suspected septicemia (quick Quick Sequential Organ Failure Assessment: respiratory rate ≥22 breaths/minute, systolic blood pressure <100 mm Hg or altered mental status with a Glasgow score < 5) ≥2
* Patients with pneumonia and [Confusion, respiratory rate ≥30 breaths/minute, blood pressure < 90/60 mm Hg, or age >65 yr.] ≥1
* Patients with very severe COPD (Forced Expiratory Volume in One Second <30%)
* Patients with COPD who have taken four or more antibiotic courses in the previous year, presence of significant bronchiectasis, and/or isolation of Pseudomonas in a previous sputum culture
* Patients with reported allergy to beta-lactams
* Patients who have taken an antibiotic in the previous two weeks
* Patients who have been hospitalized in the last two weeks
* A working diagnosis of a non-infective disorder, such as heart failure, pulmonary embolus, esophageal reflux
* Immunocompromised patients, such as HIV infection, patients taking immunosuppressive treatment, antineoplastic therapy, or systemic corticosteroids
* Currently participating in another clinical trial
* Previously participated in the STORM study
* Active neoplasia
* Terminal illness
* Institutionalized patient
* Inability/unable to understand and/or take part in the clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinical resolution | Day 14
  Number of patients with disappearance of fever, disappearance or improvement in overall condition (all scores <2), such that no additional antimicrobial treatment is necessary.

SECONDARY OUTCOMES:
Duration of antibiotic therapy | Day 14
  Number of patients discontinuing treatment in both groups and what day they discontinue recorded
Doses taken | Day 14
  Number of doses of antibiotic taken
Duration of severe symptoms | Day 14
  Number of days until the last day the patient scores 5 in any of the symptoms in the RTI diary symptom
Duration of moderate symptoms | Day 14
  Number of days until the last day the patient scores 3 in any of the symptoms in the RTI symptom diary.
Total resolution of symptoms | Day 14
  Number of days until the last day the patient scores 0 in any of the symptoms in the RTI symptom diary.
Re-attendance rate | Day 28
  Number of re-attendances to any doctor for new or worsening symptoms regarding the RTI regarding the infection
Complication rate | Day 28
  Number of complications related to the infection, such as visits to emergency departments and/or hospital admissions regarding the RTI
Absenteeism | Day 14
  Number of days of work absenteeism due to the infectious disease
Adverse events | Day 14
  Drug-associated adverse events related to the antibiotic and antibiotics changed
Use of other medication | Day 14
  Number of participants using antibiotics others than the study medication and other symptomatic therapies within the first two weeks
Health quality of life | Day 28
  Variation of the score of the health-related quality of life on days 14 and 28, compared to baseline, measured using the EuroQol instrument, including visual analogical scale, ranging from 0 (worst health condition) to 100 (best health condition)

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Morros, PhD, Study Chair — University Institute in Primary Care Research Jordi Gol, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Sharing of the individual participating data, study protocol and statistical analysis plan.
Supporting Information: Study Protocol, SAP
Time Frame: 2025 until 2027
Access Criteria: All the investigators who want to have this information shared under request.
URL: https://zenodo.org

REFERENCES:
- [Background] Llor C, Frimodt-Moller N, Miravitlles M, Kahlmeter G, Bjerrum L. Optimising antibiotic exposure by customising the duration of treatment for respiratory tract infections based on patient needs in primary care. EClinicalMedicine. 2024 Jul 3;74:102723. doi: 10.1016/j.eclinm.2024.102723. eCollection 2024 Aug. PMID 39070175
- [Derived] Morros R, Moragas A, Garcia-Sangenis A, Monfa R, Miravitlles M, Vallejo-Torres L, Jarca CI, Llor C. Tailoring Antibiotic Duration for Respiratory Tract Infections in Primary Care: Protocol for a Pragmatic Randomized Controlled Trial Study (STORM). JMIR Res Protoc. 2025 Oct 20;14:e75453. doi: 10.2196/75453. PMID 41115271